CLINICAL TRIAL: NCT06188611
Title: A Placebo Control, Randomized, Double-blind, Multicenter Phase IV Study to Investigate the Efficacy and Safety of Huazhi Rougan Granule in the Treatment of Non-alcoholic Simple Fatty Liver (Damp-heat Obstruction Syndrome: Shi-Re-Zhong-Zu Zheng)
Brief Title: A Phase IV Study of Huazhi Rougan Granule
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shandong New Time Pharmaceutical Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NTPC-HZRG-V1
Record Dates: First submitted 2023-12-13; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: A Phase IV Trial to Investigate the Efficacy and Safety of Huazhi Rougan Granule in the Treatment of Non-alcoholic Simple Fatty Liver

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Huazhi Rougan granule (Experimental): Take with boiling water ,3 times a day, for 24 weeks;
  Interventions: Drug: Huazhi Rougan Granule Placebo granule
- Placebo granule (Placebo Comparator): Take with boiling water ,3 times a day, for 24 weeks;
  Interventions: Drug: Huazhi Rougan Granule Placebo granule

INTERVENTIONS:
Drug: Huazhi Rougan Granule Placebo granule — Experimental: Huazhi Rougan granule Placebo Comparator: Placebo granule Placebo Comparator: Placebo granule

SUMMARY:
A Placebo control, Randomized, Double-blind, Multicenter Phase IV study to investigate the efficacy and safety of Huazhi Rougan granule in the treatment of non-alcoholic simple fatty liver (damp-heat obstruction syndrome: Shi-Re-Zhong-Zu Zheng)

ELIGIBILITY:
Inclusion Criteria:

* ≥18 and≤65 years old;

  * Those who meet the diagnostic criteria of non-alcoholic simple fatty liver and traditional chinese medicine syndrome classification of damp-heat obstruction syndrome;

    * Liver-to-spleen CT ratio ≤ 0.8; The imaging findings of liver were consistent with the diagnostic criteria of diffuse fatty liver; ④ Voluntarily sign informed consent. The legal representative can sign informed consent on behalf of the patient who are unable to sign； ⑤ FPG≤7.0mmol/L 、HbA1c≤6.5%；ALT、AST、TBil≤2×ULN.

Exclusion Criteria:

* Fatty liver caused by chronic heart failure, malnutrition and pregnancy, encephalopathy fatty liver syndrome (Reye syndrome), B-lipoprotein deficiency, localized fatty liver; Fatty liver caused by diabetes, long-term use of hormones, enteritis, gastrointestinal postoperative chronic infection, etc.; Small intestinal bypass surgery, hepatocyte toxicity injury, chronic febrile diseases such as tuberculosis, ulcerative nodules;；

  * Severe fatty liver with ascites, edema, hyponatremia, hypokalemia and other suspected cirrhosis; Hepatitis or cirrhosis caused by viruses, drug poisoning, immune diseases and other factors;；

    * Those who had used any Chinese or Western drugs for the treatment of simple fatty liver within one month before randomization；

      * Pregnant or lactating women, women of childbearing age who do not take effective contraceptive measures (such as condoms, hormonal contraceptives, intrauterine devices) or male subjects who do not want to use contraception;；

        * Patients with serious primary cardiovascular diseases, liver diseases, kidney diseases, hematological diseases, lung diseases, tumors, AIDS and other serious diseases that affect survival. For example: abnormal kidney function: creatinine higher than the upper limit of normal; Abnormal liver function: γ-GT>200U/L or ALT >2×ULN or AST>2×ULN; A clinically significant arrhythmia；

          ⑥ According to the 2010 guidelines for the prevention and treatment of dyslipidemia, patients with dyslipidemia requiring lipid-lowering drugs intervention：TC≥6.99mmol/L（270mg/dl）or LDL-C≥4.92mmol/L（190mg/dl）；

          ⑦ Persons without or with limited capacity for civil conduct；

          ⑧ Those who has suspected or confirmed history of alcohol abuse (alcohol equivalent male≥40g/d, female ≥20g/d) or drug abuse；

          ⑨ Allergic to the components of this drug；

          ⑩ Those who participated in other clinical investigators within 3 months prior to screening；

          ⑪ The investigators consider she/he inappropriate to participate in this study。

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2018-11-08 (Actual); Study Completion 2018-11-08 (Actual)

PRIMARY OUTCOMES:
Liver-to-spleen CT ratio | week 24

SECONDARY OUTCOMES:
Laboratory test index:Traditional Chinese medicine (TCM) syndrome points | week 24
TG、ALT、AST、γ-GT、TBIL、HOMA-IR | week 24
AE、SAE | week 24

CONTACTS AND LOCATIONS:
Locations (1):
- Longhua Hospital Shanghai University of Traditional Chinese Medicine, Shanghai, China